CLINICAL TRIAL: NCT04836208
Title: Neonatal Acquisition of ESBL-PE in a Low-income Country
Brief Title: Neonatal Acquisition of ESBL-PE in a Low-income Country - NeoLIC
Acronym: NeoLIC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Institut Pasteur (Industry)
Collaborators: Institut Pasteur de Madagascar (Other); Centre hospitalier de référence du District de Moramanga (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2020-059
Record Dates: First submitted 2021-03-31; First posted 2021-04-08 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-09

CONDITIONS: Enterobacteriaceae Infections
Keywords: new born; intra-domiciliary transmission; community; Madagascar
MeSH Terms: conditions — Enterobacteriaceae Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — * stool
  * milk for the mother of the new born
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Enterobacteriaceae, more specifically Escherichia coli and Klebsiella pneumoniae, are the bacteria most often responsible for neonatal infections in low-income countries. Infections caused by multidrug-resistant Enterobacteriaceae: Extended-spectrum beta-lactamase-producing Enterobacteriaceae (ESBL-E), are more often associated with an unfavorable outcome of the infection.

Enterobacteriaceae colonize the digestive tract which is the first step in developing a potential infection. Very few studies have been carried out at the community level. Colonization of the mother with ESBL-E is generally considered to be a major route of acquisition. The carrying of ESBL-E by other family members and other potential sources of transmission (food, objects and surfaces in contact with the newborn) have never been documented.

In addition, with a view to offering an intervention adapted to the local context, the local cultural determinants which govern the interactions of the newborn with his environment are important to understand.

DETAILED DESCRIPTION:
This is a single-center prospective cohort of all members living in the same household in which a newborn baby has just been born.

The study consists to:

* recruit a cohort of all members of 60 households in which a newborn has just been born
* carry out semi-structured interviews and direct participant observation.

This study is divided in two parts :

* the epidemiological part : the documentation of colonization by E-ESBL by sampling the stools of the newborn, of all members of the household, and sampling of food given to the child, from surfaces in contact with it.
* the anthropological part : Semi-structured interviews with key people in the structuring of the social and family environment of the newborn and participant direct observation of households.

ELIGIBILITY:
Inclusion Criteria:

1. For the epidemiological study :

   All members of 60 households in which a newborn baby has just been born

   Inclusion criteria for the mother at the time of childbirth, pregnant woman :

   _ having a monofetal pregnancy
   * residing regularly in the study area OR planning to reside in the study area during the study period;
   * having been informed of the research and collection of biological samples on herself and her newborn;
   * having given its agreement to carry out the research and the associated collection of biological samples, and;
   * having signed the informed consent (or its witness if applicable).

   Inclusion criteria for the live newborn at the time of childbirth, new born :
   * living after childbirth;
   * whose parents or legal representatives present:
   * reside regularly in the study area or plan to reside in the study area during the study period;
   * were informed of the research and the associated collection of biological samples on their newborn;
   * have given their agreement to carry out the research and the associated collection of biological samples,

   Inclusion criteria for the household member, resident:
   * from the same household as the mother-child (ren) couple included
   * Residing at least 4 nights per week in this home
   * Having given its agreement to carry out the research and the associated collection of biological samples,
   * and having signed the consent of the study (or its witness, or its legal representative if applicable)
2. for the anthropological study with interviews : 16 homes will be selected from among the 60 homes included: 8 homes in which the child has not acquired an ESBL-E during the entire follow-up and 8 homes in which the child has acquired an ESBL-E at least once during its follow-up. Among these households, interviews will be carried out with: 16 mothers or first responsible for the child in the absence of the mother 4 people with a mothering role on the child (grandmother, aunts ...) 4 minors in the families to observe 4 fathers or father figures in families to observe

   Also, interviews will be done with:

   Health actors: medical (1 midwife and 1 neighborhood doctor) and traditional (1 matron and 1 traditional practitioner from the neighborhood), 1 community health worker 1 neighborhood chief

   Inclusion criteria for semi-structured interviews :
   * people responding to the structuring functions of the child's social and family environment
   * Having given its agreement to carry out the research,
   * and having signed the consent of the study (or its witness, or its legal representative if applicable)

   For health workers and district managers, inclusion criteria for semi-structured interviews :
   * people responding to the targeted functions
   * working in the district of homes included
   * Having given its agreement to carry out the research,
   * and having signed the consent of the study (or its witness, or its legal representative if applicable)
3. For the anthropological study with observations 4 households in total among the 16 initially selected for the interviews: 2 households in which the child did not acquire ESBL-E during all the follow-up and 2 households in which the child acquired at least once an BLSE-E during his follow-up Inclusion criteria for participating direct observations

   * Residents of the same household as the mother-child (ren) couple included
   * having agreed to participate in the study
   * Having given its agreement to carry out the research,
   * and having signed the consent of the study (or its witness, or its legal representative if applicable)

Exclusion Criteria:

1. For the epidemiological part:

   * Pregnant woman: non-monofetal pregnancy
   * Newborn: died during childbirth
   * Household resident: None
2. and 3) For the anthropological part: • Semi-structured interview:

For household members:

* not responding to the structural family and social functions of the child's environment For health workers and district managers
* people not meeting the targeted functions
* not practicing in the district of homes included

  • Participant direct observation:
* Not living in the same household as the mother-child couple included

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 1. epidemiological study
     All members of 60 households in which a newborn baby has just been born
  2. anthropological study with interviews
  16 homes will be selected from among the 60 homes included: 8 homes (no ESBL-E) and 8 homes (ESBL-E). Interviews will be carried out with: 16 mothers 4 people with a mothering role on the child 4 minors in the families 4 fathers
  Also, interviews will be done with:
  Health actors: medical and traditional, 1 community health worker
  1 neighborhood chief
  3) anthropological study with observations 4 households in total among the 16 initially selected for the interviews: 2 households (no ESBL-E) and 2 households (ESBL-E)
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2021-04-30 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Number of acquisition events and the number of non-acquisition of E-ESBL in newborns for the epidemiological part | 2 years
  Identification of bacterial strains from stool and sequencing of EBSL-E strains
Number of semi-structured interviews completed for the anthropological part | 2 years
  1 or 4 hours semi-structured interviews of participants at home done by investigators
Number of participant direct observation completed for the anthropological part | 2 years
  observations of the participants at home done by investigators (2 to 4 hours in 3 to 4 sessions over 28 days)

CONTACTS AND LOCATIONS:
Overall Officials: Bich-Tram Huynh, Study Director — Institut Pasteur
Locations (1):
- Institut Pasteur de Madagascar, Antananarivo, Madagascar